CLINICAL TRIAL: NCT04903886
Title: Epidemiology of ICU-acquired Infections in Patients With Fecal Carriage of Extended Spectrum Betalactamase Enterobacteriaceae (ESBL-E)
Brief Title: Intensive Care Unit Acquired Infections in Patients Colonized With Extended Spectrum Enterobacteriaceae
Acronym: BMREA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: BMREA ( 29BRC20.0019)
Record Dates: First submitted 2021-04-28; First posted 2021-05-27 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-02

CONDITIONS: Ventilator Associated Pneumonia; Bacteremia; Abdominal Infection; Enterobacteriaceae Infections
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Bacteremia; Intraabdominal Infections; Enterobacteriaceae Infections | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All patient colonized with ESBL-E in Brest Intensive Care unit: All patient colonized with ESBL-E in Brest Intensive Care unit, in a 5 years period (2015-2019)
  Interventions: Other: observational

INTERVENTIONS:
Other: observational — observational

SUMMARY:
Worldwide emergence of extended-spectrum β-lactamase-producing Enterobacteriaceae (ESBL-E) had become a major problem in ICU, with at least 10% of incidence at the admission in Europe. A systematic rectal swab is used in 70% of French ICU to detect intestinal ESBL-E carriage The relationship between intestinal carriage and ICU-acquired infection is not perfectly known. The investigators conducted a five years study monocentric retrospective observational cohort in patients with presence of extended-spectrum β-lactamase-producing Enterobacteriaceae in systematic rectal swabs to investigate which type of infections and which bacteria are involved.

The investigators also collect data about antibiotherapy used to treat these infections.

DETAILED DESCRIPTION:
Intestinal carriage of extended-spectrum β-lactamase-producing Enterobacteriaceae (ESBL-E) had become a major problem in general population, morover in intensive care units. Systematic rectal swab for screening is done in 70% of French ICU in routine. Some studies had show a good negative predictive value of this test for ICU-acquired infection (for example ventilator-associated pneumoniae), but a poor predictive positive value. The precise relationship between intestinal carriage and ICU-acquired infection is not perfectly known.

Probabilist antibiotherapy with carbapenem for ESBL-E suspected infection are currently recommanded by national and european Guidelines, particulary in case of shock or immunodepression.

A ESBL-E systematic screening-guided strategy for probabilist antibiotherapy could be interesting, and could lead to a carbapenem or a carbapenem-sparing focused antibiotherapy.

The investigators conducted a monocentric retrospective observational cohort study in patients with presence of extended-spectrum β-lactamase-producing Enterobacteriaceae in systematic rectal swabs to investigate the number of ESBL-E related infections, the site of these infections and which species of bacteriae are involved. They also investigate which was the antibiotherapy administered, and investigate what factors lead clinicians to treat the infection with carbapenem antibiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* admitted in Brest ICU (medical or surgical)
* positive rectal swab for ESBL-Enterobacteriae screening at the admission or during the ICU stay
* written consent

Exclusion Criteria:

* refusing to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patient admitted in the ICU during a 5 years period (2015-2019) with a positive rectal swab for ESBL-Enterobacteriae screening at the admission or during the ICU stay
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
proportion of ESBL-E related infection in ICU-aquired infection | 28 days
  proportion of ESBL-E related infection in ICU-aquired infection

SECONDARY OUTCOMES:
use of carbapenem antibiotherapy | 28 days
  use of carbapenem antibiotherapy
length of ICU-stay | 28 days
  length of ICU-stay
length of hospital-stay | 28 days
  length of hospital-stay
mortality rate in ICU | 28 days
  death in ICU
mortality in hospital | 28 days
  death in hospital

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available after the publication of result and ending five years maximum following the last visit of the last patient
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. requestors will be required to sign and complete a data access agreement